CLINICAL TRIAL: NCT06413784
Title: Examining The Effect of Chronotype Differences on Sleep Quality and Pregnancy Symptoms in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10840098-772.02-6181
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Chronotype; Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: This study is a single-blind (participants), parallel trial
Who Masked: Participant
Masking Description: Participants were blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning Chronotype (Experimental): Sleep quality, gestational diabetes and pregnancy symptoms of morning chronotype individuals were examined.
  Interventions: Other: Morning chronotype
- Intermediate chronotype (Experimental): Sleep quality, gestational diabetes and pregnancy symptoms of Intermediate chronotype individuals were examined.
  Interventions: Other: Intermediate chronotype
- Evening chronotype (Experimental): Sleep quality, gestational diabetes and pregnancy symptoms of evening chronotype individuals were examined.
  Interventions: Other: Evening chronotype

INTERVENTIONS:
Other: Morning chronotype — Sleep quality, gestational diabetes and pregnancy symptoms of morning chronotype individuals were examined.
  Arms: Morning Chronotype
Other: Intermediate chronotype — Sleep quality, gestational diabetes and pregnancy symptoms of intermediate chronotype individuals were examined.
  Arms: Intermediate chronotype
Other: Evening chronotype — Sleep quality, gestational diabetes and pregnancy symptoms of evening chronotype individuals were examined.
  Arms: Evening chronotype

SUMMARY:
Purpose: The aim of this study was to examine the effect of chronotype differences on sleep quality and pregnancy symptoms in pregnant women.

Methods: Eighty-five pregnant women in the second trimester were included in the study. The chronotypes of pregnant women were determined using the Morningness-Eveningness Questionnaire (MEQ). Then, Oral Glucose Tolerance tests were performed on the participants between 24-28 weeks. Also, pregnant women's nausea and vomiting conditions with the Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) and sleep quality with Pittsburgh Sleep Quality Index (PSQI) were evaluated.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to examine the effect of chronotype differences on sleep quality and pregnancy symptoms in pregnant women.

Methods: This study is a single-blind (participants), parallel trial. It was performed in line with the principles of the Declaration of Helsinki. The followings were the study's inclusion requirements: being between the ages of 18-40, having a singleton pregnancy, being in the second trimester, and not having any known chronic disease. Exclusion criteria are working night shifts, having a high-risk pregnancy, and having a neurological or orthopedic disease. Eighty-five pregnant women in the second trimester were included in the study. The chronotypes of pregnant women were determined using the Morningness-Eveningness Questionnaire (MEQ). Then, Oral Glucose Tolerance tests were performed on the participants between 24-28 weeks. Also, pregnant women's nausea and vomiting conditions with the Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) and sleep quality with Pittsburgh Sleep Quality Index (PSQI) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-40,
* having a singleton pregnancy, being in the second trimester,
* not having any known chronic disease.

Exclusion Criteria:

* working night shifts,
* having a high-risk pregnancy,
* having a neurological or orthopedic disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The Morningness-Eveningness Questionnaire (MEQ) | 5 minutes
  It was used to measure the preference for a certain chronotype. This validated questionnaire evaluates individual differences in the degree to which respondents are aware and active at different times of the day. It has 19 items on sleep patterns and exhaustion. The responses to the scale items indicate preferences for waking and sleeping hours as well as the subjective "peak" times when respondents feel most refreshed. People were categorized as morningness chronotype (>65), intermediate chronotype (53-64), or eveningness chronotype (score of <52). The reliability of MEQ was 0.77 and the test alpha was equal to 0.78 (20).
The Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) | 5 minutes
  The PUQE is a scoring system for nausea and vomiting during pregnancy, which consists of three items. The original PUQE entailed rating the daily number of vomiting episodes, the length of nausea in hours per day, and the number of retching episodes per 12 hours. Its validation was confirmed a total score of 3-6 is considered mild nausea and vomiting, a total score of 7-12 is considered moderate nausea and vomiting, and a total score of 13-15 is considered severe nausea and vomiting
Oral Glucose Tolerance Testing (OGTT) | 15 minutes
  Pregnant women undergo a 75 g OGTT test between 24 and 28 weeks of . A plasma fasting blood glucose>126 mg/dL in a pregnant woman is considered overt diabetes (after confirmation) even if there is no prior history of diabetes. The OGTT test involves measurement of plasma glucose levels after an overnight fast (8 h), followed by oral consumption of 75 g glucose, and plasma glucose measurement at one and two hours. Gestational diabetes was defined as a fasting plasma glucose value>92 mg/dL or a one-hour plasma glucose value>180 mg/dL or a two-hour plasma glucose value>153 mg/dl.
The Pittsburgh Sleep Quality Index | 10 minutes
  It is evaluation of the sleep quality. There are 24 questions in all, 18 of which are used to determine the score. Subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disruptions, usage of sleeping pills, and dysfunction throughout the day are its seven constituent parts. The PSQI score is determined by assigning a point value between 0 and 3. A cumulative score of more than five indicates that the quality of sleep was inadequate. The score goes from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data (IPD)

REFERENCES:
- [Result] Cassidy EM, Bailey CP, Napolitano MA, Vyas AN. Sleep duration and chronotype of pregnant women in the United States: An online cross-sectional survey study. Prev Med Rep. 2022 Dec 6;31:102088. doi: 10.1016/j.pmedr.2022.102088. eCollection 2023 Feb. PMID 36820370
- See also: Sleep duration and chronotype of pregnant women in the United States: An online cross-sectional survey study. — https://pubmed.ncbi.nlm.nih.gov/36820370/